CLINICAL TRIAL: NCT00252460
Title: Evaluation of Planning Computed Tomography Scan and Magnetic Resonance Imaging Simulator Scan Co-Registration for Delineation of Gross Tumour Volume in Radiotherapy Treatment of Localized Prostate Cancer
Brief Title: CT/MRI Co-registration Prostate Cancer
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: UHN REB 03-0601-CE
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Prostatic Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Tomography, X-Ray Computed; Magnetic Resonance Imaging

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Device: Computed Tomography Scan and Magnetic Resonance Imaging

SUMMARY:
The target volume in prostate cancer radiotherapy typically consists of the entire prostate gland which is localized by contours drawn on axial computed tomography (CT) radiation planning images. Compared with CT, magnetic resonance (MR) can provide better definition of the prostate gland with respect to the surrounding tissues and the use of multi-plannar reconstruction avoids the problem of partial volume averaging inherent in CT. CT has been shown to significantly overestimate the volume of the gland using the MR-defined prostate volume as the gold standard. Co-registration of MR and CT datasets, matched on fixed bony landmarks, has enabled radiation planning using a MR-defined clinical target volumes, combined with CT-based electron density information necessary for radiation treatment planning.

Rationale and Hypothesis:

Co-registration may allow better delineation of tumour volumes in prostate cancer. This investigation is a fesibility study designed to evaluate and optimize imaging parameters and co-registration techniques for CT planning and MRI Simulator.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of Prostate Adenocarcinoma
* Undergoing RT with fiducial markers, IMRT or Escalated Dose Conformal RT

Exclusion Criteria:

* Contraindication for MRI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: prostate cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2003-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Bayley, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- University Health Network, Toronto, Ontario, Canada